CLINICAL TRIAL: NCT04878744
Title: A Feasibility Study Assessing a Green Prescription Version of a Novel App-based Intervention to Improve Wellbeing in Patients With Common Mental Health Problems
Brief Title: Feasibility Study of an App-based Intervention to Improve Wellbeing
Acronym: IWUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Derby (Other)
Responsible Party: Principal Investigator, Anna Jorgensen, Professor, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 145500
Record Dates: First submitted 2019-03-19; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: The app will be delivered as a 'green prescription' which means that health professionals will tell their patients about the intervention. If patients choose to take part, they will be allocated at random to either noticing the good things about green spaces or the good things about built spaces. This is to control for whether noticing green space or noticing other aspects of city life affects health and wellbeing. Patients will complete questionnaires about health, mental wellbeing and their feelings about nature, before, after and 3 months after using the app for one month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noticing the good things about green spaces (Experimental): The intervention condition will prompt participants once a day to notice the good things about green spaces, write notes about the 'good things in nature' and answer 4 questions about the context (e.g. were they alone or in company, exercising or passing through, did they feel comfortable in the place, what were their perceived levels of species variety).
  Participants were initially asked to use the app for one month. This was found to be associated with poor engagement at feasibility testing and so participants were asked to use the app for 7 days for the evaluation.
  Both the intervention and active control conditions are based on gratitude interventions. Practicing gratitude in controlled psychological intervention settings has been shown to have lasting effects on dispositional gratitude and psychological wellbeing (Seligman et al. 2005).
  Interventions: Behavioral: Shmapped
- Noticing the good things about built spaces (Active Comparator): In the control condition, participants will not be prompted to notice nature, rather they will be prompted to record the good things about the built environment, write notes about the 'good things in built spaces' and answer 4 questions about the context (e.g. were they alone or in company, exercising or passing through, did they feel comfortable in the place, what were their perceived levels of the area being built-up).
  Participants were initially asked to use the app for one month. This was found to be associated with poor engagement at feasibility testing and so participants were asked to use the app for 7 days for the evaluation.
  Interventions: Behavioral: Shmapped

INTERVENTIONS:
Behavioral: Shmapped — Novel app-based intervention to improve wellbeing in patients with common mental health problems.

SUMMARY:
The aim of the study is to understand how different aspects of city living affect wellbeing. The investigators hope that the results from the study will inform town planners and policy makers about how city spaces can be designed for better health and wellbeing of residents. What? This study will test the use of a new intervention amongst adults with common mental health difficulties such as depression and anxiety. The intervention will be a smartphone app which will prompt users twice a day to notice and record the good things about green spaces or built spaces around Sheffield. Previous research has shown that engaging with the natural environment can benefit health and mental wellbeing. Who? Adults over 18 years old, who have a mild to moderate common mental health problem (such as depression or anxiety), and who own a smartphone will be able to participate. Where? Participants will use the app as part of their day to day routine as they travel around Sheffield and the surrounding area. The app will prompt them to notice green or built spaces around them. How? The app will be delivered as a 'green prescription' which means that health professionals will tell their patients about the intervention. If patients choose to take part, they will be allocated at random to either noticing the good things about green spaces or the good things about built spaces. This is to control for whether noticing green space or noticing other aspects of city life affects health and wellbeing. Patients will complete questionnaires about health, mental wellbeing and their feelings about nature, before, after and 3 months after using the app for one month.

DETAILED DESCRIPTION:
The proposed feasibility study is part of a larger programme of research which asks broadly how the investigators can improve health and mental wellbeing through urban nature. The feasibility study forms part of Work Package 3 delivered by the University of Derby. The main study in work package 3 will recruit over 1,000 Sheffield residents to evaluate an app-based intervention to improve wellbeing through prompting people to notice the good things about nature. For the feasibility study, the investigators will pilot a green prescription version of this intervention with 100 adults who have common mental health difficulties. The feasibility study asks the question of how feasible it is to recruit patients to the study using a green prescription method of clinician signposting (measured through referral numbers and referral source). It also asks whether there are any health and mental wellbeing benefits to adults with common mental health problems (measured through health and mental wellbeing questionnaires completed at pre, post and 3 months follow-up).

People who are exposed to nature, or feel connected with it, present higher levels of general health and subjective wellbeing. Individuals with mental health problems have been shown to particularly benefit from nature-based interventions . In a recent Natural England report, evidence from a range of nature-based interventions for mental health patients and found the following benefits: i) reduced depression and anxiety; ii) increased positive affect; iii) increased social contact; and iv) increased mental wellbeing.

At present, the knowledge about the beneficial effects of nature is insufficient to be applied in a systematic way in health promotion and urban planning. There is a need to move beyond cross-sectional evidence and natural experiments. Work package 3 aims to fill this research gap through a largescale controlled study, which will employ a robust quasi-experimental methodology to look at the health and wellbeing benefits of engaging the public with urban nature. To go beyond cross-sectional data, the study will randomise participants to an app-based intervention which will either prompt them to notice the good things about green spaces or to an active control condition which will prompt them to notice the good things about built spaces.

As part of work package 3 the investigators will conduct a feasibility study assessing a green prescription version of the app-based intervention for adults with common mental health problems. This will help estimate the wider potential for using the nature-based intervention in a clinical population. 'The natural environment has potential to offer cost-effective solutions to address health inequalities and produce positive physical and mental health outcomes'. Some of the data collected will be used to estimate QALYs and to look at cost utility of the intervention in this group of patients.

The research proposal was developed by the principal investigator (Prof. Anna Jorgensen, Sheffield University) and collaborators from Sheffield University, Derby University and Herriot-Watt University. The team is multidisciplinary encompassing public health, landscape, architecture and design, psychology and mental health, and economics. Internal peer-review was sought from experts in this field of research before submitting the research bid and the bid was reviewed and approved for funding by the Natural Environment Research Council.

Input into study design has also come from an advisory panel which includes several clinicians, one of whom has expertise in green prescriptions and social prescribing (Dr William Bird) and stakeholders (e.g. The Wildlife Trust, TCV Green Gyms and the Centre for Sustainable Healthcare). Stakeholders and community groups have also given us feedback on the project at a project launch meeting and those of whom provided contact details to stay involved, have been contacted and consulted about the green prescription. The investigators have costed into the grant to have patient and public involvement in the app development. The Recovery Enterprise (a Sheffield-based mental health organisation) will provide feedback on the design and usability of the app and will be involved in field-testing of the app with us.

Recruitment For the recruitment strategy the investigators have consulted with the clinicians on the advisory panel (Dr Liz Walton & Dr William Bird), and with Sheffield-based GPs, CCG, and IAPT professionals and third sector organisations offering green prescriptions or social prescriptions. The investigators have also taken guidance from two recently published Natural England reports on the topics of nature-based interventions for mental health care and good practice in social prescribing for mental health.

The investigators will be asking Sheffield-based GPs, IAPT clinicians and third sector organisations (such as People Keeping Well, Voluntary Action Sheffield, The Recovery Enterprise and Flourish) to signpost eligible participants to the study website via posters, leaflets and brief discussions about the study. Participants who are interested in taking part will be signposted to the study website where they can read more about the research aims and the app-based intervention. A copy of the participant information and consent sheet is available on the study website and on the app itself. Contact details for the lead researcher are available should participants have any further questions. For transparency about what data will be collected, why it will be collected and how it will be processed and stored, the investigators have written a privacy impact assessment (as recommended by the ICO guidance on mobile app security) and this is available to view from the website (http://iwun.uk/).

If participants decide they would like to take part, they can download the app onto their phone where they will again be presented with the information and consent sheet, and study instructions. Participants will consent by tapping 'yes I consent' on their phone. This is a standard procedure for obtaining consent in similar app-based research studies. It is made clear to participants in the information sheet that if they change their mind about participating, they can withdraw from the study without giving a reason and can withdraw their data anytime before the 1st of January 2018.

Consent the investigators will be asking Sheffield-based GPs, IAPT clinicians and third sector organisations (such as People Keeping Well, Voluntary Action Sheffield, The Recovery Enterprise and Flourish) to signpost eligible participants to the study website via posters, leaflets and brief discussions about the study. Participants who are interested in taking part will be signposted to the study website where they can read more about the research aims and the app-based intervention. A copy of the participant information and consent sheet is available on the study website and on the app itself. Contact details for the lead researcher are available should participants have any further questions.

Participants will be asked to indicate that they consent to participate in the study by tapping 'I agree' in the app. This comes after reading the full participant information sheet. By clicking "I agree" participants confirm that:

* They are at least 18 years old
* They know what information they'll be sending to us, why the investigators are collecting it, and what the investigators will use the information for
* They agree to send this data to us
* They agree to us getting and storing information about their geographical location using GPS
* They understand participants can leave the study at any time
* This is their mobile device

Participants will be able to review the information sheet at any time either in the app by clicking the 'About' option in the menu, or on the study website (http://iwun.uk/). The information sheet details what the study is about, who can take part, what is involved in taking part and how long it will take, what data will be collected (including information collected using the phone sensors), what will happen to the data, information about confidentiality, anonymity, withdrawal, and who to contact if participants have further questions. For transparency about what data will be collected, why it will be collected and how it will be processed and stored, the investigators have written a privacy impact assessment (as recommended by the ICO guidance on mobile app security) and this is available to view from the website (http://iwun.uk/).

Risks, burdens and benefits The main risk to participants is securely storing their anonymised data. The investigators are aware of risks to data held on smartphones through previous literature. The investigators have taken advice from the app developers, the UK Data Centre and have read the guidance document from the ICO on the best procedures for storing app data securely. This is as follows: Data in the phone will be secured using the normal phone's methods (password, digital fingerprints, etc.). Access will happen through the unique identifier provided by Google and Apple (e.g. Google and password or a Sheffield mapping app password) so the data collected will only be accessible by the right owner. Through these procedures the investigators will reduce the risk of data being accessed by third parties.

Measures will be taken to prevent location data being misused. The frequency of location data collection is the minimum necessary to answer the research questions about exposure to green and built spaces. Location will be tagged by the app i)every 30 minutes; ii)when participants enter and exit a publicly accessible green or built space; and iii)to prompt participants to notice nature/built environment as they enter an area of green space/grey space (predefined by geofences provided by work package 1). For a selection of more prominent city green spaces the investigators may also ask participants permission via the app if the investigators can track their location as they move through the park (every 20 seconds). This will allow some case study analysis of what particular green space features (e.g. woodland, grassland etc) participants tend to be drawn to. The participant will decide the duration to allow prompts to be sent in when they set-up the app. Participants movements outside their selected hours will not be tracked. In this way the investigators are collecting the minimum data on participant location to allow the study questions to be answered. This allows us to analyse which environments are most beneficial to health and wellbeing.

The investigators have a written contract between (University of Derby) and the app developers (Furthermore) to ensure that data protection requirements for the study are met. Information about the study, data collection, storage and who to contact for further information will always be available to participants through the app and the study website. The investigators also have a privacy impact assessment which the investigators have shared with the app developers, the database custodians (Derby University) and participants via the website. All researchers and app developers have undergone data security training with the University of Sheffield and researchers handling personal data have up to date GCP training and DBS clearance. Participants will be allocated at random to either the intervention condition of noticing the good things about nature or the control condition of noticing the good things about built spaces. The investigators expect both of these conditions to be beneficial to wellbeing as they both get participants to notice and reflect upon the good things in their surroundings. However, the investigators do expect noticing green spaces to have a greater beneficial effect given previous literature.

The information sheet informs participants that the data collected are confidential and anonymous. The investigators are not collecting any personal data (i.e. data that would allow the identification of that person)other than ethnicity. The investigators are collecting the minimum required data to answer the research questions.

The privacy impact assessment details what data will be collected, why it is being collected (with justification from previous literature) and how the data will be processed and stored. This is available to participants through the study website.

Principle 1 - Justify the purpose(s) for obtaining the information. The research question asks whether urban nature can improve health and wellbeing, and asks what type of natural environments provide the greatest benefit. Hence the investigators will collect questionnaire data on health (EQ5D) and wellbeing (Recovering quality of life scale-ReQoL & Types of positive affect scale-TPAs). Two of these scales (EQ5d & ReQoL) will also be used to estimate QALYs and conduct a cost utility analysis. To assess whether the app is having the desired intention of increasing engagement with the natural environment, the investigators will measure nature connectedness (Nature connectedness scale & single item Inclusion of Self in Nature scale). These questionnaires will be completed at pre, post and 3 months follow-up to using the app.

The app will prompt participants once a day to notice and record the good things about green spaces or built spaces. As part of the intervention participants write notes about these good things at the end of each day. Participants are given the choice of allowing the app to track their location every 30 minutes during the day and whenever they enter and exit a publicly accessible green or built space. This provides data to answer the research question about what exposure participants have to green or built space during their day and which type of natural or built environments provide the greatest wellbeing benefits.

When participants enter their daily notes they will be asked 4 questions about context e.g. were they alone or with others, were they exercising or simply walking through a place, how did they feel about that place, what was the variety of species like. These contextual influences have been shown to act as moderators between accessing green spaces and wellbeing. Hence these items will be used in analyses to assess the context in which wellbeing benefits are gained. Other potential moderators will be asked at baseline, these include age, gender, ethnicity, postcode (1st 4 digits only), access to a garden and previous connection with nature.

The tracking data is potentially quite sensitive data which is why the investigators have taken advice from several app developers (who are experienced in this type of app that uses tracking) about how to collect and securely store this data. The investigators have also taken advice from the UK Data Centre and have followed guidance from the Information Commissioners Office (ICO) document 'Privacy in mobile apps: Guidance for app developers'. The investigators have chosen to collect the minimum tracking data to answer the study questions. Geofences of publicly accessible green and built spaces will be programmed into the app. As participants pass through these geofences the app will record their location. This will give us an estimate of their exposure to green and built spaces throughout the day and allow prompts to occur when the participant is in a green or built space. When a participant then walks near to one of these geofences the phone will prompt them to notice the green or built space around them. The app will also record participants location every 30 minutes to gain information about general exposure to indoors/outdoors and green/built space throughout daylight hours.

Principle 2 - The investigators will not collect any person-identifiable data in this study. None of the demographics data collected, or the participants partial postcode are enough alone or necessarily in combination to identify an individual with any certainty. Tracking data can be sensitive and so the investigators are only collecting the minimum location tracking data to answer the study questions. Ethnicity data is deemed personal by the Data Protection Act and will therefore be stored in a separate database to the remainder of the data and will be linked for analysis using an anonymised linking ID code.

Principle 3 - See principle 2. The investigators will not collect any person-identifiable data and any sensitive data such as ethnicity, will be held in a separate database to other data.

Principle 4 - See principles 2 & 3.

Principle 5 - The investigators are not collecting any person identifiable data. A data protection plan has been written by the researchers and this forms part of the contract between the researchers and the app developers. The investigators have also written a privacy impact assessment which has been shared with the app developers, database custodians (Derby University) and participants via the study website. The researchers and app developers have undertaken data security training with the University of Sheffield and the lead researcher has valid GCP certificates and has applied for basic DBS clearance.

Principle 6 - The investigators are aware of risks to data held on smartphones through previous literature. The investigators have taken advice from the app developers, the data protection act 1998, the UK Data Centre and an ICO guidance document on the best procedures for storing mobile app data securely. The investigators will not be collecting any identifiable data or tissue samples. The investigators will conform with Article 8 of the European Human Rights Convention ensuring that the collected and processed information will not be used by a public authority to interfere in the private life of a person unless this is necessary for national security or public safety. In such a case, The investigators will comply with the duty of having to alert public authorities to the ethical and practical implications of the research results. Conflict of interest The lead researcher in this study and the study team are all researchers/lecturers and not healthcare professionals. There is no conflict of interest in this research.

At the end of the study participants will be sent a debriefing statement via the app. This will thank participants for their participation, give further information of the studies aims, provide information about where the results from the study can be found and details of any public dissemination events, provide contact details for the lead researcher, and inform participants that they can delete the app from their smartphone if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Having a mild to moderate common mental health problem (such as depression and/or anxiety)
* Owning a smartphone

Exclusion Criteria:

* Aged under 18 years old
* Do not have a mild to moderate common mental health problem (depression and/or anxiety)
* Do not own a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Number of participants completing the study | post-intervention at 1 month
  Whether the participant remains in the study until post-intervention measures
Number of participants who write daily notes | post-intervention at 1 month
  Whether the participant engages with the app at least 50% of the time by writing notes about the good things they noticed when prompted daily by the app.
Change in Recovering Quality of Life scale (Brazier et al., 2014) from baseline to post-intervention | Baseline and post-intervention at 1 month
  This is a mental health specific quality of life scale. Possible scores range from 0-40, with higher scores indicating greater quality of life.
Change in Inclusion of self in nature scale (Schultz, 2001) between baseline and post-intervention | Baseline and post-intervention at 1 month
  This is a single item measure of connection to nature. Scores range from 0-100 with higher scores indicating greater nature connection.
Change in Types of positive affect scale (Gilbert et al., 2009) between baseline and post-intervention | Baseline and post-intervention at 1 month
  This scale measures activated and relaxed constructs of positive affect. Higher scores indicate greater positive affect. There are three subscales of Relaxed positive affect (scores range 0-48), Safe positive affect (scores range 0-32) and Activated positive affect (scores range 0-32).
Change in Nature Relatedness scale (Nisbet & Zelenski 2008) between baseline and post-intervention | Baseline and post-intervention at 1 month
  This is a measure of connection to nature. Scores range from 1-30 with higher scores indicating greater nature connection.
Change in Engagement with Natural Beauty scale (Diessner et al. 2008) between baseline and post-intervention | Baseline and post-intervention at 1 month
  This is a measure of noticing natures beauty. Scores range from 1-28, with higher scores indicating greater appreciation of natures beauty.
Change in EQ-5D-European Quality of Life scale (Rabin, 2001) between baseline and post-intervention | Baseline and post-intervention at 1 month
  This is a measure of physical and mental wellbeing. Questions are scored individually and there are four questions. Lower scores indicate better health, so a maximum score of 1 per question indicates optimal health. There is also a visual analogue scale scored 0-100 with 100 indicating the best health score.
Details about participants visit to green/built spaces | post-intervention at 1 month
  4 single questions ask about 1) the variety of wildlife or how built-up the area was (responses are none or lots, 2) how that place made them feel (participants respond by clicking a smiley face or a sad face), 3)who they were with (response options include no one, friends/family/partner, Coworker/course mate, in a crowd, pet or other) , and 4) what they were doing (response options include walking, exercising, relaxing, travelling, other).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators will not collect any person-identifiable data in this study. None of the demographics data collected, or the participants partial postcode are enough alone or necessarily in combination to identify an individual with any certainty. Tracking data can be sensitive and so the investigators are only collecting the minimum location tracking data to answer the study questions. Ethnicity data is deemed personal by the Data Protection Act and will therefore be stored in a separate database to the remainder of the data and will be linked for analysis using an anonymised linking ID code.
  Research participants' self-assessed health and wellbeing and perceptions of the natural environment (urban parks and green spaces) will be shared with other researchers via the UK Data Service at the end of the project.
Supporting Information: Study Protocol
Time Frame: Data will be available from 5th June 2019